CLINICAL TRIAL: NCT02450552
Title: A Phase 2 Pharmacodynamic Trial of Ezogabine (Retigabine) on Neuronal Excitability in Amyotrophic Lateral Sclerosis
Brief Title: Clinical Trial of Ezogabine (Retigabine) in ALS Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brian Wainger (Other)
Collaborators: ALS Association (Other); GlaxoSmithKline (Industry); Harvard University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Brian Wainger, Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014D002776
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Lou Gehrig
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral ezogabine 600 mg/day (Experimental)
  Interventions: Drug: Ezogabine
- Oral ezogabine 900 mg/day (Experimental)
  Interventions: Drug: Ezogabine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezogabine — Potiga is FDA-approved for adjunctive treatment of partial-onset seizures in patients aged 18 years and older who have responded inadequately to several alternative treatments.
  Other Names: Potiga; Retigabine
  Arms: Oral ezogabine 600 mg/day; Oral ezogabine 900 mg/day
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
This study evaluates the effect of retigabine (600 mg/day, 900 mg/day, or placebo) on motor neuron activity in people with Amyotrophic Lateral Sclerosis (ALS). The total study duration is approximately 14 weeks. ALS subjects will take study drug for approximately 10 weeks.

DETAILED DESCRIPTION:
One of the major disease features of ALS is the progressive death of motor neurons. Human, rodent and stem cell-based model studies support the hypothesis that neuronal hyperexcitability may contribute to neurodegeneration in both sporadic and familial ALS. The investigators are doing this research study to find out whether retigabine will reduce motor neuron excitability in people with ALS. the investigators will also determine whether the drug is tolerable and safe for patients with ALS.

The proposed study will determine how the potassium channel opener ezogabine (retigabine) affects neurophysiological measures of upper and lower motor neuron excitability in ALS patients as assessed by transcranial magnetic stimulation (TMS) and threshold tracking nerve conduction studies (TTNCS), respectively. The study will include the recruitment of approximately 60 unmatched healthy control subjects for analysis of variability of the neurophysiological tests prior to recruitment of ALS subjects. There will also be 12 matched healthy control subjects, recruited at the same time as ALS subjects.

ELIGIBILITY:
ALS Subject Inclusion Criteria:

* Male or female, aged 18 to 80.
* Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria.
* Slow vital capacity (SVC) measure ≥ 50% of predicted for gender, height and age at the Screening Visit,OR in the opinion of the SI, ability to perform and safely complete all study visit procedures.
* Subjects must not have taken riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days prior to the Screening Visit and continue on the stable dose throughout the course of the study (riluzole-naïve subjects are permitted in the study).
* Subjects must be able to swallow oral medication at the Screening Visit and expected to be able to swallow tablets throughout the course of the study.
* Capable of providing informed consent and following trial procedures.
* Geographically accessible to the site.
* Women must not be able to become pregnant (e.g., post menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and three months after study completion. Adequate contraception includes: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal contraception, for example patch or contraceptive ring), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.
* Use of medications known to affect the neurophysiology measures in the study must be scheduled, not as needed (pro re nata, PRN). A subject must have been on a fixed dose for 30 days prior to the Screening Visit, and there must be no reason to believe that a subsequent change would be necessary during the course of the study. These medications include: benzodiazepines, muscle relaxants, tricyclic antidepressants, selective serotonin reuptake inhibitors, non-selective serotonin reuptake inhibitors, hypnotics (including anti-histamines) and anti-cholinergics.
* TMS shows sufficient MEP amplitude and/or NCS studies show sufficient CMAP amplitude.

ALS Subject Exclusion Criteria:

* Medical condition, laboratory finding, or physical exam finding that precludes participation.
* Serum AST and ALT value >2.0 times the upper normal limit
* Clinically significant conduction abnormalities on electrocardiogram or a known history of cardiac arrhythmia, myocardial infarction within the past 24 months, or congestive heart failure.
* Estimated glomerular filtration rate < 50 mL/min at Screening Visit.
* Concomitant digoxin treatment.
* Known allergic reactions to components of the study product(s).
* Exposure to any other agent currently under investigation for the treatment of patients with ALS (off-label use or investigational) within 30 days of the Screening Visit including ezogabine, exposure to cell replacement therapy within six months of the Screening Visit or any prior intraparenchymal cell replacement injection within the spinal cord or brain at anytime in the past.
* Presence of tracheostomy at the Screening Visit.
* History of clinically significant urinary retention, , or current use of medications to treat urinary retention.
* History of drug and or alcohol abuse within 12 months of the Screening Visit.
* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, according to SI judgment.
* Clinically significant history of unstable or severe cardiac, oncologic, hepatic, or renal disease, or other uncontrolled medical condition.
* Presence of feeding tube.
* Current use of antipsychotic, antiepileptic (except benzodiazepines, gabapentin, pregabalin) or class 1 (e.g. flecainide) or class 3 (e.g. amiodarone) antiarrhythmic medications. Quinidine or a quinidine-containing drug is allowed if the quinidine dose is not greater than 20 mg/day (for a full list of medications, please reference the study MOP).
* Inability to perform either TMS or NCS studies due to insufficient MEP or CMAP amplitude.
* Pregnant women or women currently breastfeeding.
* Contraindication to TMS studies including ferromagnetic metal in the head or neck (potentially found in aneurysm clips, implanted medication pumps, implanted brain stimulators, pacemakers, cochlear implants), or history of epilepsy. Dental fillings are permitted.
* Anything else that, in the opinion of the SI, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.

Healthy Control Subject Inclusion Criteria:

* Male or female, aged 18 to 80.
* Absence of a known neurological disorder.
* Capable of providing informed consent and following trial procedures.
* Geographically accessible to the site.
* Age (+/- 10 years and site-matched to a ALS participant within 6 months of their Baseline visit).[Matched controls only]
* TMS shows sufficient MEP amplitude and/or NCS studies show sufficient CMAP amplitude (amplitudes defined in MOP).
* Use of medications known to affect the neurophysiology measures in the study must be scheduled, not as needed (pro re nata, PRN). A subject must have been on a fixed dose for 30 days prior to the Screening Visit, and there must be no reason to believe that a subsequent change would be necessary during the course of the study. These medications include: benzodiazepines, muscle relaxants, tricyclic antidepressants, selective serotonin reuptake inhibitors, non-selective serotonin reuptake inhibitors, hypnotics (including anti-histamines) and anti-cholinergics.

Healthy Control Subject Exclusion Criteria:

* History of ALS or other neurodegenerative disease.
* Presence of positive family history of ALS.
* Current use of an antipsychotic or antiarrhythmic medication
* Definitely or possibly pregnant.
* Contraindication to TMS studies including ferromagnetic metal in the head or neck ( potentially found in aneurysm clips, implanted medication pumps, implanted brain stimulators, pacemakers, cochlear implants), or history of epilepsy. Dental fillings are permitted.
* Anything that, in the opinion of the SI, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-06; Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Wainger, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (12):
- United States (12):
  - Barrow Neuological Institute, Phoenix, Arizona
  - Cedars-Sinai, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Augusta University (Georgia Regents Medical Center), Augusta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Hospital for Special Surgery, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Penn State College of Medicine Milton S. Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Derived] Wainger BJ, Macklin EA, Vucic S, McIlduff CE, Paganoni S, Maragakis NJ, Bedlack R, Goyal NA, Rutkove SB, Lange DJ, Rivner MH, Goutman SA, Ladha SS, Mauricio EA, Baloh RH, Simmons Z, Pothier L, Kassis SB, La T, Hall M, Evora A, Klements D, Hurtado A, Pereira JD, Koh J, Celnik PA, Chaudhry V, Gable K, Juel VC, Phielipp N, Marei A, Rosenquist P, Meehan S, Oskarsson B, Lewis RA, Kaur D, Kiskinis E, Woolf CJ, Eggan K, Weiss MD, Berry JD, David WS, Davila-Perez P, Camprodon JA, Pascual-Leone A, Kiernan MC, Shefner JM, Atassi N, Cudkowicz ME. Effect of Ezogabine on Cortical and Spinal Motor Neuron Excitability in Amyotrophic Lateral Sclerosis: A Randomized Clinical Trial. JAMA Neurol. 2021 Feb 1;78(2):186-196. doi: 10.1001/jamaneurol.2020.4300. PMID 33226425

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Started | 19 | 23 | 23
Completed | 14 | 23 | 18
Not Completed | 5 | 0 | 5
Not completed — Withdrawal by Subject | 4 | 0 | 4
Not completed — Physician Decision | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo | Total
Number analyzed (Participants) | 19 | 23 | 23 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.91 (9.10) | 57.4 (8.01) | 58.1 (9.55) | 58.34 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 4 | 20
  Male | 13 | 13 | 19 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 22 | 22 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 17 | 23 | 23 | 63
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 23 | 23 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Short-interval Intracortical Inhibition (SICI) Measured by Transcranial Magnetic Stimulation (TMS)
Description: Short-interval intracortical inhibition (SICI) or paired-pulse SICI is defined as the ratio of the response after a conditioning pulse equal to 80% of resting motor threshold (RMT) is administered 3 ms prior to the signaling pulse divided by motor evoked potential (MEP) amplitude. Transcranial magnetic stimulation (TMS) is a neurophysiologic test for assessing upper motor neuron function. Change in SICI will be assessed by transcranial magnetic stimulation (TMS) after treatment with 900 mg/day or 600 mg/day of ezogabine vs. matched oral placebo.
Time Frame: Screening, Baseline, Week 6, Week 8
Population: As a result of electrophysiologic response, good quality data was defined based on the central reader's evaluation.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
Unitless
  Screening: number analyzed (Participants) | 12 | 11 | 13
  Screening | 1.180 (1.108) | 0.965 (1.302) | 0.784 (0.560)
  Baseline: number analyzed (Participants) | 13 | 16 | 13
  Baseline | 1.347 (1.662) | 0.952 (1.138) | 0.755 (0.539)
  Week 6: number analyzed (Participants) | 9 | 12 | 14
  Week 6 | 1.100 (1.066) | 0.675 (0.613) | 0.777 (0.442)
  Week 8: number analyzed (Participants) | 8 | 10 | 15
  Week 8 | 0.948 (1.169) | 0.617 (0.455) | 0.834 (0.488)

2. Secondary Outcome: Change in Resting Motor Evoked Potential (MEP) Threshold (Prespecified Secondary Outcome of Primary Importance)
Description: Resting Motor Evoked Potential (MEP) is the magnetic field strength, measured as a percentage of the maximum stimulator output, that produces at least a 0.05 mV response in at least 5 of 10 consecutive trials.Change in resting MEP threshold will be assessed by Transcranial Magnetic Stimulation (TMS).
Time Frame: Screening, Baseline, Week 6, Week 8
Population: Data of low quality may have been removed from the number of participants analyzed based on the central reader's evaluation.
Measure: Mean (Standard Deviation); unit: percentage of the maximum output
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
percentage of the maximum output
  Screening: number analyzed (Participants) | 12 | 11 | 13
  Screening | 51.250 (14.379) | 52.000 (11.480) | 56.308 (13.804)
  Baseline: number analyzed (Participants) | 13 | 16 | 13
  Baseline | 48.385 (14.373) | 54.250 (11.018) | 57.231 (13.498)
  Week 6: number analyzed (Participants) | 9 | 12 | 14
  Week 6 | 50.111 (14.066) | 57.583 (15.365) | 54.714 (12.313)
  Week 8: number analyzed (Participants) | 8 | 10 | 14
  Week 8 | 46.00 (10.876) | 56.700 (13.039) | 55.357 (10.149)

3. Secondary Outcome: Change in MEP Amplitude
Description: Motor Evoked Potential (MEP) amplitude is defined as the response when a stimulus equal to 120% of Resting Motor Threshold (RMT) is administered. MEP amplitude is calculated as the geometric mean of replicate estimates. Change in MEP will be assessed by Transcranial Magnetic Stimulation (TMS).
Time Frame: Screening, Baseline, Week 6, Week 8
Population: Data of low quality were removed from analysis as a result of the central reader's evaluation standards.
Measure: Geometric Mean (Standard Deviation); unit: Millivolts
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
Millivolts
  Screening: number analyzed (Participants) | 12 | 11 | 13
  Screening | 0.639 (0.635) | 1.210 (1.958) | 0.845 (0.626)
  Baseline: number analyzed (Participants) | 13 | 16 | 13
  Baseline | 0.395 (0.282) | 0.954 (1.402) | 1.098 (1.197)
  Week 6: number analyzed (Participants) | 9 | 12 | 14
  Week 6 | 1.78 (1.568) | 0.914 (0.861) | 0.454 (0.339)
  Week 8: number analyzed (Participants) | 8 | 10 | 14
  Week 8 | 0.571 (0.345) | 1.129 (0.600) | 0.450 (0.299)

4. Secondary Outcome: Change in Duration of Cortical Silent Period
Description: Cortical silent period (CSP) is the suppression of voluntary muscle contraction elicited by stimulation equal to 120% of resting motor threshold (RMT). CSP duration is measured from the time of the muscle activity suppression to return of muscle activity. Change in duration of cortical silent period is assessed by Transcranial Magnetic Stimulation (TMS).
Time Frame: Screening, Baseline, Week 6, Week 8
Population: Data of low quality were removed from analysis population as a result of the central reader's evaluation standards.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
Milliseconds
  Screening: number analyzed (Participants) | 12 | 11 | 13
  Screening | 99.542 (39.153) | 69.273 (29.921) | 88.831 (39.519)
  Baseline: number analyzed (Participants) | 13 | 16 | 13
  Baseline | 80.223 (23.440) | 76.006 (30.459) | 80.638 (32.894)
  Week 6: number analyzed (Participants) | 9 | 12 | 14
  Week 6 | 96.844 (43.426) | 74.917 (36.338) | 83.479 (32.920)
  Week 8: number analyzed (Participants) | 8 | 10 | 14
  Week 8 | 88.000 (32.258) | 58.870 (21761) | 87.479 (39.839)

5. Secondary Outcome: Change in Intracortical Facilitation
Description: Paired-pulse Intracortical facilitation (ICF) is defined as the ratio of the response after a conditioning pulse equal to 80% of Resting Motor Threshold (RMT) is administered 15 milliseconds prior to the signaling pulse divided by Motor Evoked Potential (MEP) amplitude. ICF is calculated as the geometric mean of replicate estimates. Change in intracortical facilitation is assessed by Transcranial Magnetic Stimulation (TMS).
Time Frame: Screening, Baseline, Week 6, Week 8
Population: Data of low quality were removed from analysis population as a result of the central reader's evaluation standards.
Measure: Geometric Mean (Standard Deviation); unit: Unitless
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
Unitless
  Screening: number analyzed (Participants) | 13 | 11 | 13
  Screening | 1.829 (0.862) | 1.849 (1.669) | 1.653 (0.907)
  Baseline: number analyzed (Participants) | 13 | 16 | 13
  Baseline | 2.420 (2.356) | 2.073 (2.075) | 1.531 (0.906)
  Week 6: number analyzed (Participants) | 9 | 12 | 14
  Week 6 | 1.894 (1.177) | 1.535 (1.472) | 1.571 (1.298)
  Week 8: number analyzed (Participants) | 8 | 10 | 14
  Week 8 | 1.779 (1.627) | 1.466 (0.836) | 1.514 (0.817)

6. Secondary Outcome: Change in Electrotonus
Description: Change in depolarizing electrotonus at 90 to 100 milliseconds was assessed by threshold tracking axonal nerve conduction studies (TTNCS). TTNCS is a neurophysiologic test for assessing lower motor neuron function.
Time Frame: Screening, Baseline, Week 6, Week 8
Population: Data of low quality were removed from analysis population as a result of the central reader's evaluation standards.
Measure: Mean (Standard Deviation); unit: percentage of threshold
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
percentage of threshold
  Screening: number analyzed (Participants) | 14 | 18 | 21
  Screening | 52.275 (14.924) | 48.144 (8.636) | 44.532 (6.666)
  Baseline: number analyzed (Participants) | 14 | 19 | 18
  Baseline | 46.278 (7.663) | 48.901 (9.327) | 46.574 (6.689)
  Week 6: number analyzed (Participants) | 10 | 13 | 18
  Week 6 | 50.187 (6.645) | 51.857 (7.303) | 44.898 (6.082)
  Week 8: number analyzed (Participants) | 7 | 12 | 16
  Week 8 | 50.108 (2.533) | 48.552 (13.422) | 47.010 (6.212)

7. Secondary Outcome: Change in Strength Duration Time Constant
Description: Assessed by threshold tracking axonal nerve conduction studies (TTNCS).
Time Frame: Screening, Baseline, Week 6, Week 8
Population: Data of low quality were removed from analysis population as a result of the central reader's evaluation standards.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
Milliseconds
  Screening: number analyzed (Participants) | 14 | 18 | 20
  Screening | 0.521 (0.084) | 0.451 (0.096) | 0.505 (0.086)
  Baseline: number analyzed (Participants) | 14 | 20 | 19
  Baseline | 0.522 (0.084) | 0.454 (0.084) | 0.488 (0.078)
  Week 6: number analyzed (Participants) | 10 | 13 | 19
  Week 6 | 0.416 (0.141) | 0.480 (0.165) | 0.546 (0.120)
  Week 8: number analyzed (Participants) | 7 | 13 | 16
  Week 8 | 0.341 (0.079) | 0.461 (0.134) | 0.497 (0.173)

8. Secondary Outcome: Change in Recovery Cycle
Description: Lower motor neuron excitability can be measured using change in recovery cycle of superexcitability. Change in recovery cycle of superexcitability after first pre-pulse is assessed by threshold tracking axonal nerve conduction studies (TTNCS). Threshold-tracking nerve conduction studies is a neurophysiologic test for assessing lower motor neuron function.
Time Frame: Screening, Baseline, Week 6, Week 8
Population: Data of low quality were removed from analysis as a result of the central reader's evaluation standards.
Measure: Mean (Standard Deviation); unit: percentage of threshold
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
percentage of threshold
  Screening: number analyzed (Participants) | 14 | 18 | 20
  Screening | -30.45 (8.694) | -28.12 (8.401) | -27.77 (7.955)
  Baseline: number analyzed (Participants) | 13 | 19 | 19
  Baseline | -31.39 (6.896) | -27.40 (6.993) | -28.16 (7.589)
  Week 6: number analyzed (Participants) | 9 | 12 | 18
  Week 6 | -37.59 (5.066) | -37.48 (7.451) | -28.37 (7.835)
  Week 8: number analyzed (Participants) | 5 | 12 | 15
  Week 8 | -38.20 (4.965) | -33.15 (13.874) | -29.26 (5.880)

9. Secondary Outcome: Muscle Cramping Frequency
Description: Frequency of muscle cramping and maximum pain from muscle cramping was collected by subjects via self-report using a daily muscle cramping diary.
Time Frame: Week 1 through Week 10
Population: Discrepancies in the number of subjects analyzed are a result of subjects with missed data collection during the specific time points.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
Days
  Week 1: number analyzed (Participants) | 17 | 21 | 22
  Week 1 | 12.176 (15.233) | 8.738 (14.477) | 9.536 (15.909)
  Week 2: number analyzed (Participants) | 17 | 20 | 22
  Week 2 | 9.235 (11.729) | 7.083 (11.558) | 8.273 (10.968)
  Week 3: number analyzed (Participants) | 17 | 20 | 22
  Week 3 | 10.906 (13.532) | 7.750 (12.268) | 10.170 (13.915)
  Week 4: number analyzed (Participants) | 17 | 20 | 22
  Week 4 | 12.018 (18.824) | 9.135 (12.664) | 106.19 (14.016)
  Week 5: number analyzed (Participants) | 15 | 17 | 22
  Week 5 | 12.533 (15.824) | 10.265 (13.404) | 8.955 (13.268)
  Week 6: number analyzed (Participants) | 15 | 15 | 23
  Week 6 | 11.033 (11.705) | 8.333 (10.887) | 8.539 (10.869)
  Week 7: number analyzed (Participants) | 15 | 14 | 23
  Week 7 | 9.400 (10.716) | 9.714 (12.755) | 9.609 (12.551)
  Week 8: number analyzed (Participants) | 15 | 15 | 22
  Week 8 | 11.211 (13.521) | 9.067 (11.151) | 9.282 (12.244)
  Week 9: number analyzed (Participants) | 14 | 15 | 21
  Week 9 | 12.786 (14.154) | 9.933 (11.750) | 11.190 (16.162)
  Week 10: number analyzed (Participants) | 14 | 16 | 20
  Week 10 | 13.179 (14.953) | 10.188 (12.296) | 13.600 (16.162)

10. Secondary Outcome: Hand Held Dynamometry Force Measurement for Abductor Pollicis Brevis
Description: Hand held dynamometry (HHD) will be used as a quantitative measure of muscle strength of the abductor pollicis brevis (APB) muscle. HHD will be self-report by study participants using a daily muscle cramping diary.
Time Frame: Screening, Baseline, Week 4, Week 6, Week 8, Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
kilograms (kg)
  Screening: number analyzed (Participants) | 19 | 22 | 21
  Screening | 6.721 (4.548) | 8.577 (6.927) | 7.448 (4.048)
  Baseline: number analyzed (Participants) | 19 | 22 | 22
  Baseline | 6.584 (4.022) | 6.641 (4.901) | 7.164 (4.716)
  Week 4: number analyzed (Participants) | 18 | 21 | 22
  Week 4 | 6.461 (4.002) | 7.333 (5.839) | 6.686 (5.115)
  Week 6: number analyzed (Participants) | 16 | 19 | 22
  Week 6 | 6.838 (3.569) | 6.921 (5.570) | 6.300 (5.167)
  Week 8: number analyzed (Participants) | 13 | 18 | 22
  Week 8 | 7.015 (4.398) | 5.633 (4.015) | 6.523 (4.523)
  Week 12: number analyzed (Participants) | 15 | 18 | 21
  Week 12 | 5.887 (3.696) | 5.439 (3.609) | 5.643 (4.523)

11. Secondary Outcome: Proportion of Days With Fasciculations
Description: For the purpose of this study, a fasciculation is a brief, spontaneous contraction affecting a small number of muscle fibers, often causing a flicker of movement under the skin. Defining interference with daily activities may be different for each subject and defining daily activities will be different for each subject. Subjects will self report by diary, days with fasciculations.
Time Frame: Week 1 through Week 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Proportion of Days
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
Proportion of Days
  Week 1: number analyzed (Participants) | 14 | 13 | 14
  Week 1 | 0.918 (0.134) | 0.659 (0.415) | 0.745 (0.368)
  Week 2: number analyzed (Participants) | 14 | 13 | 14
  Week 2 | 0.918 (0.229) | 0.637 (0.435) | 0.776 (0.325)
  Week 3: number analyzed (Participants) | 14 | 13 | 14
  Week 3 | 0.796 (0.366) | 0.648 (0.439) | 0.816 (0.334)
  Week 4: number analyzed (Participants) | 14 | 13 | 14
  Week 4 | 0.752 (0.352) | 0.637 (0.450) | 0.806 (0.348)
  Week 5: number analyzed (Participants) | 13 | 13 | 15
  Week 5 | 0.879 (0.285) | 0.659 (0.461) | 0.733 (0.374)
  Week 6: number analyzed (Participants) | 13 | 11 | 14
  Week 6 | 0.868 (0.288) | 0.714 (0.438) | 0.765 (0.418)
  Week 7: number analyzed (Participants) | 13 | 10 | 14
  Week 7 | 0.912 (0.277) | 0.767 (0.417) | 0.786 (0.379)
  Week 8: number analyzed (Participants) | 13 | 11 | 15
  Week 8 | 0.868 (0.294) | 0.688 (0.460) | 0.714 (0.432)
  Week 9: number analyzed (Participants) | 12 | 10 | 14
  Week 9 | 0.893 (0.293) | 0.657 (0.472) | 0.857 (0.296)
  Week 10: number analyzed (Participants) | 12 | 10 | 13
  Week 10 | 0.869 (0.319) | 0.700 (0.483) | 0.813 (0.380)

12. Secondary Outcome: Number of Participants Who Tolerate Study Drug
Description: Participants will be judged tolerant of study drug if they reached their target dose and remain on study drug until planned discontinuation. Tolerability will be summarized as the proportion of participants in a treatment group who are tolerant of study drug.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
Number analyzed (Participants) | 19 | 23 | 23
Participants | 14 | 11 | 23

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the date the first subject signed consent, November 30, 2015, to the date the last subject completed the last study visit, February 27, 2018, a total of about 2 years, 3 months.
Arm/Group | Oral Ezogabine 900 mg/Day | Oral Ezogabine 600 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/23 | 0/23
Other Adverse Events (participants affected / at risk) | 19/19 | 23/23 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Ezogabine 900 mg/Day (N=19) | Oral Ezogabine 600 mg/Day (N=23) | Placebo (N=23)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed Level of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Ezogabine 900 mg/Day (N=19) | Oral Ezogabine 600 mg/Day (N=23) | Placebo (N=23)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (6) | 3 (3)
Paraesthesia Oral (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0)
Tongue Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (3) | 0 (0)
Fatigue (General disorders) | 7 (7) | 11 (12) | 6 (6)
Gait Disturbance (General disorders) | 2 (2) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 7 (7) | 4 (7)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bacterial Test (Investigations) | 1 (1) | 0 (0) | 0 (0)
Crystal Urine Present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 5 (6)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 3 (4)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Balance Disorder (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 1 (2) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 8 (9) | 5 (6) | 3 (3)
Dysarthria (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Dysstasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (3) | 5 (6)
Language Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Contractions Involuntary (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 7 (7) | 2 (2) | 1 (1)
Speech Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (3) | 1 (2) | 0 (0)
Euphoric Mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination, Visual (Psychiatric disorders) | 4 (5) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Perseveration (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Urinary Hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 4 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 0 (0)
Increased Viscosity Of Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (5) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hypersecretion (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT02450552/SAP_000.pdf
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/52/NCT02450552/Prot_001.pdf